CLINICAL TRIAL: NCT01752933
Title: A Phase 2 Study of SGI-110 in the Treatment of Advanced Hepatocellular Carcinoma (HCC) Subjects Who Failed Prior Treatment With Sorafenib
Brief Title: SGI-110 in the Treatment of Advanced Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGI-110-03
Record Dates: First submitted 2012-12-17; First posted 2012-12-19 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SGI-110 (Experimental): SGI-110 administered subcutaneously (SC) daily on Days 1 - 5 every 28 days
  Interventions: Drug: SGI-110

INTERVENTIONS:
Drug: SGI-110 — SGI-110 will be administered by subcutaneously (SC) on Days 1 - 5 every 28 days until disease progression or unacceptable toxicity

SUMMARY:
A Phase 2 open-label, single-arm, non-randomized study in the treatment of advanced hepatocellular carcinoma (HCC) patients who failed prior treatment with sorafenib using a Simon's 2-stage design. A set minimum number of patients must demonstrate disease control at 16 weeks to proceed to Stage 2. At Stage 2, a set number of patients must have disease control at 16 weeks to declare that SGI-110 is of interest in the treatment of advanced HCC after failure of prior sorafenib.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Histological or cytological confirmed hepatocellular carcinoma with advanced stage disease
3. Received prior sorafenib treatment, and showed evidence of disease progression, which is defined as Investigator verified radiologic progression, or intolerance of prior systemic therapy, which is defined as having had clinically significant adverse events that persisted despite one or more dose reductions or interruptions
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
5. Acceptable organ function
6. Signed an approved informed consent

Exclusion Criteria:

1. Known hypersensitivity to SGI-110
2. Adequate washout of prior radiation, chemotherapy or other locoregional therapy
3. Abnormal left ventricular ejection fraction
4. Uncontrolled ischemic heart disease or a history of congestive cardiac failure
5. Known brain metastases
6. Clinically evident ascites
7. Child-Pugh C cirrhosis or Child-Pugh B cirrhosis with more than 7 points
8. Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, non-metastatic prostate cancer with normal prostate-specific antigen (PSA) or other cancer from which the subject has been disease free for at least three years
9. Known history of human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (15):
  - City of Hope National Medical Center, Duarte, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Northwestern University: Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Louisville James Graham Brown Cancer Center, Louisville, Kentucky
  - Columbia University Medical Center - Herbert Irving Comprehensive Cancer Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Hollings Cancer Center, Charleston, South Carolina
  - The Jones Clinic, PC, Germantown, Tennessee
  - Mary Crowley Medical Research Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - UW Carbone Cancer Center, Madison, Wisconsin
- Canada (5):
  - University of British Columbia and Vancouver General Hospital, Vancouver, British Columbia
  - The Ottawa Hospital Cancer Center, Ottawa, Ontario
  - Sunnybrook HealthScience Centre, Toronto, Ontario
  - CHUM Hopital St-Luc, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- United Kingdom (4):
  - University of Liverpool Clatterbridge Cancer Center, Liverpool
  - Cambridge University Hospitals NHS Foundation Trust, London
  - Imperial College Healthcare NHS Foundation Trust, London
  - University College London, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 68 patients were screened for enrollment in the study. Of these, 16 were screen failures. Reasons for screen failure included not meeting all eligibility criteria (14 patients) and withdrawal of consent (2 patients).
Pre-assignment Details: Of the 52 patients enrolled in the study, 2 did not receive any treatment. Reasons for not receiving treatment included death for one patient and no longer meeting eligibility criteria for the second patient.
Groups:
- Guadecitabine 60 mg/m^2: Guadecitabine (SGI-110) 60 mg/m^2 subcutaneously (SC) on Days 1 - 5 of each 28-day cycle
- Guadecitabine 45 mg/m^2: Guadecitabine (SGI-110) 45 mg/m^2 SC on Days 1 - 5 of each 28-day cycle
Period: Treatment
Arm/Group | Guadecitabine 60 mg/m^2 | Guadecitabine 45 mg/m^2
Started ("Reason Not Completed" shown below are reasons for treatment discontinuation) | 4 (Includes all patients who received any treatment) | 46 (Includes all patients who received any treatment)
Completed (Treatment continued as long as patient was benefitting from treatment with manageable side effects) | 0 (Completion not applicable for this survival study) | 0 (Completion not applicable for this survival study)
Not Completed | 4 | 46
Not completed — Disease Progression | 3 | 29
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Adverse Event | 1 | 4
Not completed — Physician Decision | 0 | 3
Not completed — Death | 0 | 2
Not completed — Hepatocellular carcinoma not confirmed | 0 | 1
Not completed — Patient noncompliant | 0 | 1
Not completed — Patient unable to travel to appointments | 0 | 1
Period: Overall Study and Follow-up
Arm/Group | Guadecitabine 60 mg/m^2 | Guadecitabine 45 mg/m^2
Started ("Reason Not Completed" shown below are reasons for study discontinuation) | 4 (Includes all patients who received any treatment) | 46 (Includes all patients who received any treatment)
Completed | 0 (Completion not applicable for this survival study) | 0 (Completion not applicable for this survival study)
Not Completed | 4 | 46
Not completed — Death | 4 | 34
Not completed — Sponsor terminated study/Database lock | 0 | 7
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: The total number of subjects presented for Baseline Analysis (50 subjects) is less than the total presented in Participant Flow (52 subjects) because 2 subjects were withdrawn from the study prior to receiving treatment and thus were not assigned to a treatment group.
Groups:
- Guadecitabine 60 mg/m^2: Guadecitabine (SGI-110) 60 mg/m^2 SC on Days 1 - 5 of each 28-day cycle
- Total: Total of all reporting groups
Arm/Group | Guadecitabine 60 mg/m^2 | Guadecitabine 45 mg/m^2 | Total
Number analyzed (Participants) | 4 | 46 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 33 | 37
  >=65 years | 0 | 13 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 7 | 7
  Male | 4 | 39 | 43
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 7 | 7
  United States | 4 | 39 | 43

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR) at 16 Weeks for Patients Treated With Guadecitabine After Failure of Sorafenib
Description: Percentage of patients achieving a best overall response of complete response (CR) or partial response (PR) plus subjects with stable disease at 16 weeks after the start of treatment. Response was assessed based on the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for target and non-target lesions using computed tomography (CT) or magnetic resonance imaging (MRI) as follows: Complete Response (CR), disappearance of all target lesions, disappearance of all non-target lesions, and normalization of tumor marker level; Partial Response (PR), at least a 30% decrease in the sum of diameters of target lesions from baseline; Progressive Disease (PD), at least a 20% relative increase and 5 mm absolute increase in the sum of diameters of target lesions, and unequivocal progression of non-target lesions; Stable Disease, neither sufficient shrinkage to quality for PR nor sufficient increase to qualify for PD (Eisenhauer et al. 2009, Eur. J. Cancer 45:228-247).
Time Frame: 16 weeks
Population: Patients who met major inclusion/exclusion criteria and followed the study protocol without a significant deviation (1 patient excluded because did not have confirmed HCC; 4 patients excluded because did not have a Week 16 assessment).
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Guadecitabine 45 mg/m^2: Guadecitabine (SGI-110) 45 mg/m^2 on Days 1 - 5 of each 28-day cycle
Arm/Group | Guadecitabine 60 mg/m^2 | Guadecitabine 45 mg/m^2
Number analyzed (Participants) | 4 | 41
percentage of patients | 25.0 [0.6 to 80.6] | 24.4 [12.4 to 40.3]

2. Secondary Outcome: Safety and Tolerability of Guadecitabine
Description: Number of patients with serious adverse events and adverse events
Time Frame: Varied by patient (median number of treatment cycles was 2.0 (range 2-8) in 60 mg/m^2 group, and 4.0 (range 1-13) in 45 mg/m^2 group
Population: Includes all patients who received any guadecitabine
Measure: Count of Participants; unit: Participants
Arm/Group | Guadecitabine 60 mg/m^2 | Guadecitabine 45 mg/m^2
Number analyzed (Participants) | 4 | 46
Participants
  Serious Adverse Event | 1 | 21
  Adverse Event | 4 | 46

3. Secondary Outcome: Alpha Fetoprotein Response as a Result of Guadecitabine Administration
Description: Percentage of patients with best post baseline alpha fetoprotein reduction of 50% or more
Time Frame: as for outcome 2
Population: Includes all patients who received any guadecitabine
Measure: Count of Participants; unit: Participants
Arm/Group | Guadecitabine 60 mg/m^2 | Guadecitabine 45 mg/m^2
Number analyzed (Participants) | 4 | 46
Participants | 0 | 2

4. Secondary Outcome: Duration of Response
Description: Duration of response as measured in days. Included subjects with a complete response or partial response based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: From time of first response until disease progression or date of death due to any cause, whichever occurred earlier; an average of 192 days.
Population: Assessed for patients who had a clinical response
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Guadecitabine 60 mg/m^2 | Guadecitabine 45 mg/m^2
Number analyzed (Participants) | 1 | 10
days | 262 | 144 [109.0 to 240.0]

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival measured in days. Progression-free survival was defined as the time interval from the date of the first dose of study treatment to the earlier of 1) documented radiologic progression per RECIST v1.1 or clinical progression, or 2) death due to any cause.
Time Frame: Through completion of response assessments (i.e., until disease progression or treatment discontinuation), an average of 112 days.
Population: Includes all patients who received any guadecitabine
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Guadecitabine 60 mg/m^2 | Guadecitabine 45 mg/m^2
Number analyzed (Participants) | 4 | 46
days | 55 [50.0 to 262.0] | 82.5 [57.0 to 113.0]

6. Secondary Outcome: Overall Survival
Description: Overall survival measured in days.
Time Frame: Through completion of study survival follow-up, an average of 270 days.
Population: Includes all patients who received any guadecitabine
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Guadecitabine 60 mg/m^2 | Guadecitabine 45 mg/m^2
Number analyzed (Participants) | 4 | 46
days | 294 [103.0 to 683.0] | 245 [148.0 to 303.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events included events that first occurred or worsened after the first dose of study drug until 30 days after the last dose of study drug or the start of alternative anticancer treatment for HCC, whichever occurred first. Events that occurred more than 30 days after the last dose of study treatment or start of alternative cancer treatment were also considered treatment emergent if they were both serious and related to treatment.
Arm/Group | Guadecitabine 60 mg/m^2 | Guadecitabine 45 mg/m^2
All-Cause Mortality (participants affected / at risk) | 4/4 | 34/46
Serious Adverse Events (participants affected / at risk) | 1/4 | 21/46
Other Adverse Events (participants affected / at risk) | 4/4 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guadecitabine 60 mg/m^2 (N=4) | Guadecitabine 45 mg/m^2 (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 5
Atrial fibrillation (Cardiac disorders) | 0 | 1
Adrenal haemorrhage (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Blood creatinine increased (Investigations) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Guadecitabine 60 mg/m^2 (N=4) | Guadecitabine 45 mg/m^2 (N=46)
Anaemia (Blood and lymphatic system disorders) | 1 | 11
Leukopenia (Blood and lymphatic system disorders) | 1 | 21
Lymphopenia (Blood and lymphatic system disorders) | 0 | 10
Neutropenia (Blood and lymphatic system disorders) | 4 | 39
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 20
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 7
Abdominal pain (Gastrointestinal disorders) | 1 | 8
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4
Ascites (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 11
Diarrhoea (Gastrointestinal disorders) | 2 | 11
Nausea (Gastrointestinal disorders) | 2 | 11
Stomatitis (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 9
Chills (General disorders) | 0 | 5
Early satiety (General disorders) | 0 | 3
Fatigue (General disorders) | 3 | 24
Injection site erythema (General disorders) | 2 | 3
Injection site haematoma (General disorders) | 1 | 3
Injection site pain (General disorders) | 2 | 21
Injection site reaction (General disorders) | 0 | 6
Mucosal inflammation (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 1 | 9
Pyrexia (General disorders) | 1 | 9
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 5
Urinary tract infection (Infections and infestations) | 0 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 8
Aspartate aminotransferase increased (Investigations) | 1 | 14
Blood alkaline phosphatase increased (Investigations) | 1 | 10
Blood bilirubin increased (Investigations) | 0 | 4
Hypoalbuminemia (Investigations) | 0 | 3
Weight decreased (Investigations) | 0 | 4
Weight increased (Investigations) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5
Dizziness (Nervous system disorders) | 1 | 6
Dysgeusia (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 2 | 6
Neuropathy peripheral (Nervous system disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 1 | 4
Mental status changes (Psychiatric disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 5
Hypertension (Vascular disorders) | 0 | 8
Hypotension (Vascular disorders) | 0 | 5
Atrial fibrillation (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 1
Gingival swelling (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 1
Injection site induration (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The original starting dose of 60 mg/m^2 guadecitabine was reduced to 45 mg/m^2 after dose-limiting toxicities occurred in the first 4 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No